CLINICAL TRIAL: NCT00163696
Title: Measurements of Inhomogeneity of the Small Airway With Patients With Cystic Fibrosis, Asthma and Bronchiolitis Obliterans Syndrome (Post Transplant) Using the Multi Breath Nitrogen Washout Technique
Brief Title: Multi Breath Nitrogen Washout (MBNW) as a Measure of Small Airway Function in Patients With Respiratory Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: The Alfred (Other)
Other Study IDs: MBNW alfred
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2007-07-26 (Estimated); Status verified 2005-09

CONDITIONS: Cystic Fibrosis; Asthma; Bronchiolitis Obliterans; Lung Transplantation
Keywords: MBNW; Ventilation; small airways; Lung Transplant recipients (Bronchiolitis Obliterans syndrome)
MeSH Terms: conditions — Cystic Fibrosis; Asthma; Bronchiolitis Obliterans; Respiratory Aspiration; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The researchers are investigating a novel technique, the multi breath nitrogen washout technique, to measure airway changes in various respiratory diseases.

DETAILED DESCRIPTION:
It is well documented that there are significant ventilatory changes in respiratory diseases such as cystic fibrosis, asthma and the onset of bronchiolitis obliterans syndrome (BOS) following chronic rejection of lung transplantation. At present, we use measures such as spirometry and lung biopsies to determine the changes of airway function and disease severity. Our aim is to develop a novel technique called the multi breath nitrogen washout (MBNW) which we believe is able to measure the inhomogeneity of ventilation in both the larger airways (conductive region, generation 1 - 16) as well as the smaller airways (acinar region 17 - 23). Our belief is that these measurements are much more subtle than current techniques and will be more sensitive in measuring large and small airway changes in disease. The MBNW can also give us an insight as to which particular zones of the lung are affected in differing respiratory disease. For example, it is believed that BOS begins at the distal portion of the lung (acinar region) and proceeds towards the proximal zone (conductive). However, at present no current techniques can differentiate between damage to the acinar zone and the conductive zone or indeed accurately measure small airway (acinar zone) function. We believe the the MBNW has the capacity to do so.

ELIGIBILITY:
Inclusion Criteria:

* Doctor diagnosed cystic fibrosis, asthma
* Lung transplant recipient

Exclusion Criteria:

* Smoke history of less than 10 pack years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Thompson, Principal Investigator — Head of Physiology Services, Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia